CLINICAL TRIAL: NCT05970211
Title: Early Age-Related Hearing Loss Investigation Pilot Study
Acronym: P-EARLHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Michelle Arnold, Assistant Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005599
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hearing Intervention Group (Experimental): Adults aged 55-75 with hearing loss who have little/no prior experience with hearing aids will be enrolled in the hearing intervention group.
  Interventions: Device: Phonak Audeo Lumity Receiver in Canal Hearing Aid

INTERVENTIONS:
Device: Phonak Audeo Lumity Receiver in Canal Hearing Aid — bilateral receiver in canal hearing aids provided as part of a best practices hearing loss intervention including devices, hearing centered counseling, and self management skills training for hearing loss

SUMMARY:
The purpose of this clinical trial pilot is to obtain feasibility and pilot data necessary to inform the hearing intervention being designed for a larger R01 clinical trial that seeks to determine whether best practice hearing aid intervention impacts hearing-related outcomes in adults with hearing loss aged 55 to 75 years.

Secondary purposes include: To determine what effects best practice hearing aid intervention has on physical, social, and quality of life outcomes in adults with hearing loss aged 55 to 75 years.

DETAILED DESCRIPTION:
This is an observational pre-post intervention feasibility study. In addition to the objective finding that adults with hearing loss experience higher rates of cognitive decline, they also tend to report lesser degrees of physical activity and increased cognitive fatigue, which is the feeling of tiredness or having a lack of energy. Unfortunately, the mechanism by which hearing loss relates to physical activity and fatigue, and the effect of hearing aids as an intervention to improve these factors, is unclear. Thus, the purpose of this study is twofold: First, we will establish the feasibility of administering a best practices hearing aid intervention to a sample of adults from the target age range of 55 - 75 years old to inform the larger clinical trial; Second, we will collect pilot data to explore the relationships between hearing loss, physical activity, socialization, fatigue and hearing-related outcomes before and after hearing aid intervention.

There are no experimental or investigational devices or agents used in this study. We are providing best-practices standard of care hearing intervention including hearing aids. We are additionally tracking activity using the ActiGraph wGT3X-BT, an FDA-approved Class II medical device that tracks continuous, high resolution physical activity and sleep/wake information.

Participation involves a minimum of 6 in-office study visits. Intervention sessions occur approximately 2 weeks apart, with a final long-term outcome session occurring approximately 6-months post the baseline intervention session.

Significant others of participants are invited to join the study and contribute data related to their own quality of life and their observations of the effects of the hearing intervention on the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 to 75 years old with little or no experience with hearing aids
* English or Spanish speakers

Exclusion Criteria:

* Unable to complete written questionnaires on a tablet without assistance
* Refer for cognitive screening score based on criteria using the Mini Mental State Examination

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Objective Physical Activity | 2-week measurement taken between 4- and 6- months post study enrollment
  Activity level as measured by research-grade accelerometer

SECONDARY OUTCOMES:
Words in Noise Test | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Measures speech perception in noise performance
International Outcome Inventory for Comprehensive Hearing Intervention | Measured at 6-months post study enrollment
  Self-reported hearing aid benefit measure
Client Oriented Scale of Improvement | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported hearing aid benefit measure
Hearing Handicap Inventory for Adults | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported hearing handicap
Center for Epidemiological Studies Depression and Hopelessness Scale | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported depression
Speech, Spatial and Qualities of Hearing Scale | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported hearing difficulties
Social Network Index | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported social network information
UCLA Loneliness Scale | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported loneliness
The Positive and Negative Affect Schedule | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported positive and negative affect/mood
The World Health Organization Well-Being Index | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported well being
The Vanderbilt Fatigue Scale for Adults | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported fatigue
Research & Development Short Form Survey (RAND36) | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported quality of life
Single-item sedentary questionnaire | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported physical activity
Modified four-square step test | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Measures physical function
Expanded short physical performance battery | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Measures lower extremity function
Baecke Physical Activity Questionnaire | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported physical activity
PROMIS v2.0 Mobility Questionnaire | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported mobility
User Experience Questionnaire+ | Measured at time of study enrollment; between 6- and 8-weeks post study enrollment; and at 6-months post study enrollment
  Self-reported hearing device user experience

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States